CLINICAL TRIAL: NCT03943082
Title: A Pilot Feasibility Study for Improving Patient Access to Cancer Clinical Trials (iMPACT): A Financial Reimbursement Program for Patients in Cancer Therapeutic Clinical Trials
Brief Title: Impact of Phone Call About Financial Reimbursement Program on Access to Cancer Clinical Trials
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual for Feasibility Met
Sponsor: University of California, San Francisco (Other)
Collaborators: Lazarex Cancer Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 189819; NCI-2019-00171 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Malignant Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms | interventions — Aftercare; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A : Usual Care (FRP Only) (Active Comparator): Patients or parents/legal guardians of patients receive FRP brochure at the time of iMPACT consent.
  Interventions: Behavioral: Cancer Educational Materials; Behavioral: Questionnaire
- Cohort A: Usual Care + Intervention (FRP + Follow-up) (Experimental): Patients or parents/legal guardians of patients receive FRP brochure at the time of iMPACT consent and a follow-up phone call on day 3 after iMPACT consent.
  Interventions: Behavioral: Cancer Educational Materials; Other: Follow-Up Care; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Cancer Educational Materials — Receive FRP brochure
Other: Follow-Up Care — Receive follow-up phone call
  Arms: Cohort A: Usual Care + Intervention (FRP + Follow-up)
Behavioral: Questionnaire — Ancillary studies
  Other Names: Questionnaires

SUMMARY:
This trial studies how well a follow-up phone call regarding financial reimbursement program (FRP) works in improving cancer patients' access to therapeutic cancer clinical trials. Follow-up phone call intervention regarding FRP may improve recruitment of cancer patients to cancer therapeutic clinical trials.

DETAILED DESCRIPTION:
There are limited financial models that address the economic hardship associated with clinical research participation and how it might restrict clinical research access. The Lazarex Foundation offers a financial reimbursement program (FRP) to help patients and caregivers cover the out-of-pocket costs associated with clinical trial participation for almost ten years.

iMPACT is a pilot study to assess the overall feasibility of conducting a multi-center trial of the Lazarex sliding scale FRP among sociodemographically diverse patients of all cancer types enrolling/potentially enrolling in therapeutic clinical trials (TCTs). The study will formalize informing patients or parents/legal guardians of patients about the Lazarex sliding-scale FRP in order to evaluate whether operationalizing intensive follow-up about the Lazarex FRP improves recruitment to cancer TCTs.

All patients or parents/legal guardians of patients will be offered information about the FRP at initial time of TCT discussion/consent for the iMPACT study, however, participants will be randomized 1:1 to receive an additional follow-up call about the FRP or no follow-up call (usual care). Participants who are randomized to usual care will be provided a phone number for the Lazarex Foundation that they or their parent or legal guardian may contact directly. Therefore all patients or parents/legal guardians of patients in the study have access to FRP eligibility assessment through the Lazarex Foundation.

Participants or parents/legal guardians of participants will be surveyed at baseline (time of consent to iMPACT) and interviewed 30 days after consent to iMPACT. If a participant enrolls in a therapeutic clinical trial, he/she will also be given an additional survey after TCT participation and interviewed up to 90 days after TCT participation.

ELIGIBILITY:
Inclusion Criteria:

COHORT A:

* Eligible patients to be randomized for the iMPACT study must:

  1. Carry a diagnosis of cancer
  2. Patient is considered potentially eligible for a cancer therapeutic clinical trial (TCT) and is being offered an opportunity to sign an informed consent document for the cancer TCT
* Eligible patients to receive FRP (these documents will be requested by Lazarex Foundation, however research coordinator at site can help patient collect documents):

  1. Have a household income =< 700% of the 2018 Health and Human Services (HHS) Poverty Guidelines
  2. Willing to provide proof of household income. Acceptable proof of income documents are: first two pages of signed copy of income tax return, or if a return is not filed, a copy of the most recent pay stub, unemployment check, Supplemental Security Income (SSI), Social Security Disability (SSD), or public assistance benefit notification. If a patient is not employed, they must submit a signed letter stating their current financial situation

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who sign consent to improving Patient Access to Cancer Clinical Trials (iMPACT) study among patients who are offered enrollment | Up to 90 days after therapeutic clinical trial (TCT) participation
  The point estimate and 95% confidence interval (CI) of the proportion will be obtained within each site, furthermore, by cancer type and by phase of the clinical trial within each site.

SECONDARY OUTCOMES:
Proportion of patients who sign consent for cancer TCT as well as by cancer type and phase of clinical trial within each arm | At day 30
  Two-sample proportion test between two arms will be used between two arms within each site. The point estimate and 95% confidence interval (CI) of the proportion will be obtained within each site by cancer type and by phase of the clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Borno, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No